CLINICAL TRIAL: NCT06589076
Title: Correlation of Apical Periodontitis With Anxiety and Depression: A University Case-Control Study
Brief Title: Apical Periodontitis and Mental Health
Status: Active, not recruiting | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Simone Grandini, Professore, University of Siena
Other Study IDs: MHAP001
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Apical Periodontitis; Anxiety; Depression
Keywords: Oral Health; Mental Health; Apical Periodontitis; Anxiety; depression; smokers
MeSH Terms: conditions — Periapical Periodontitis; Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group (AP+):: This group consists of participants who have apical periodontitis (AP), an oral inflammatory condition. These participants are diagnosed with AP based on radiographic evidence. They may exhibit symptoms of AP, but AP is often asymptomatic, so radiographic confirmation is key.
  Interventions: Diagnostic Test: Clinical and Radiographic assessment + Questionnaires
- Control Group (AP-):: This group consists of participants who do not have apical periodontitis (AP). These participants are healthy individuals with no clinical or radiographic signs of apical periodontitis. They will be matched with the case group based on age, gender, and other relevant characteristics, but they will not have any dental lesions related to apical periodontitis.
  Interventions: Diagnostic Test: Clinical and Radiographic assessment + Questionnaires

INTERVENTIONS:
Diagnostic Test: Clinical and Radiographic assessment + Questionnaires — * Clinical and radiographic examination to assess oral health and apical periodontitis.
  * Questionnaires to assess Anxiety and depression.

SUMMARY:
This study is investigating the relationship between anxiety, depression and apical periodontitis (AP), a common oral inflammatory condition. The research is being conducted at the Unit of Endodontic and Conservative Dentistry, University of Siena, Italy, with participants aged over 18. Participants are divided into two groups: those with apical periodontitis and those without. The study aims to determine whether there is an association between anxiety, depression (assessed using the Hamilton Anxiety/Depression Rating Scale), and the presence or severity of apical periodontitis. Data collection includes dental exams, radiographs, and anxiety and depression assessments. This research may help to better understand how mental health and dental health are connected.

DETAILED DESCRIPTION:
The aim of the present case-control study is to evaluate the association between apical periodontitis (AP) and mental health conditions, specifically anxiety and depression. Subjects will be enrolled from the Unit of Endodontics and Conservative Dentistry of the University of Siena.

The inclusion criteria of the study are healthy patients older than 18 years, the ability and willingness to give informed consent, and the presence of untreated periapical lesions for the case group. Participants without apical periodontitis will be included in the control group. Participants affected by systemic diseases such as diabetes or rheumatoid arthritis, those using corticosteroid drugs, and those in stage 3 or 4 of periodontitis will be excluded. Additional exclusion criteria include the use of antibiotics within the last 6 months, inability to give informed consent, and pregnancy or lactation.

Seventy-one subjects fulfilling the described criteria will be enrolled and allocated into two distinct groups based on the presence or absence of apical periodontitis. Group 1 will consist of patients with radiographic evidence of AP, and Group 2 will consist of healthy controls free from clinical and radiographic signs of AP. The AP+ group will include patients with at least one tooth showing radiographic evidence of apical radiolucency.

To perform the initial screening, participants will undergo panoramic radiography, clinical examination, and periapical radiographs using the long cone paralleling technique to assess suspected AP. The following parameters will be recorded:

* The number of decayed, missing, and filled teeth (DMFT index)
* The number of teeth with apical periodontitis
* Periapical Index (PAI) Score

All mental health assessments will be conducted using standardized psychiatric scales, including the Hamilton Depression Rating Scale (HAM-D) and the Hamilton Anxiety Rating Scale (HAM-A), to evaluate the severity of depression and anxiety, respectively.

Additionally, smoking status (current, former, or non-smoker) will be recorded to explore its association with apical periodontitis and its potential impact on anxiety and depression scores.

The results expected from this study are:

* A potential correlation between apical periodontitis and increased anxiety and depression scores (HAM-A and HAM-D).
* A possible association between smoking habits and the severity of mental health conditions in relation to apical periodontitis.

This study may help to elucidate the connection between oral and mental health, highlighting the importance of holistic health care approaches that consider both physical and psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to give written consent;
* Age above 18 years old;
* Presence of an untreated periapical lesion for the case group;
* Absence of a periapical lesion for the control group.

Exclusion Criteria:

* Diabetes;
* Rheumatoid Arthritis;
* Use of corticosteroid drugs;
* Stage 3 and 4 of periodontitis;
* Inability or unwillingness to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants fulfilling the previously described inclusion criteria will be allocated into two distinct groups based on the presence or absence of apical periodontitis (AP). Group 1 will consist of 36 patients showing radiographic signs of apical periodontitis (AP+), while Group 2 will include 35 healthy individuals (AP-) with no clinical or radiographic evidence of AP, serving as controls. Participants in both groups will be matched based on age, sex, and other relevant characteristics. AP cases will be defined as patients with at least one tooth exhibiting radiographic evidence of apical radiolucency, graded using Peri Apical Index (PAI) Score.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) Score | At baseline (during participant enrollment and evaluation)
  The severity of anxiety symptoms is measured using the Hamilton Anxiety Rating Scale (HAM-A). This scale assesses both psychological (mental distress) and somatic (physical symptoms) aspects of anxiety. Scores range from 0 to 56, with higher scores indicating more severe anxiety. The association between HAM-A scores and the presence of apical periodontitis (AP) will be analyzed.
Hamilton Depression Rating Scale (HAM-D) Score | At baseline (during participant enrollment and evaluation)
  The severity of depression is assessed using the 17-item Hamilton Depression Rating Scale (HAM-D). The scale evaluates a range of depressive symptoms such as mood disturbances, guilt, insomnia, anxiety, and somatic concerns. Scores range from 0 to 52, with higher scores indicating more severe depression. The association between HAM-D scores and the presence of apical periodontitis (AP) will be analyzed.
Periapical Index (PAI) Score | At baseline (during participant enrollment and evaluation)
  The Periapical Index (PAI) score is used to assess the severity of apical periodontitis. The score ranges from 1 to 5, with higher scores indicating more severe periapical inflammation. The association between PAI scores and anxiety (HAM-A) and depression (HAM-D) scores will be analyzed.

SECONDARY OUTCOMES:
Decayed, Missing, and Filled Teeth (DMFT) Index | At baseline (during participant enrollment and evaluation)
  The DMFT index is recorded to evaluate the overall dental health of participants. It assesses the number of decayed, missing, and filled teeth, providing a comprehensive measure of oral health. The association between DMFT index and anxiety (HAM-A) and depression (HAM-D) scores will be analyzed.
Smoking Status and Its Association with Mental Health and Oral Health | At baseline (during participant enrollment and evaluation)
  Smoking status (current smoker, former smoker, non-smoker) will be assessed to evaluate its relationship with apical periodontitis and its impact on depression (HAM-D) and anxiety (HAM-A) scores. The analysis will explore whether smoking is a confounding factor in the association between mental health and oral health conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Grandini, PhD, DDS, Principal Investigator — University of Siena
Locations (1):
- Azienda Ospedaliera Universitaria Senese, Siena, Tuscany, Italy